CLINICAL TRIAL: NCT05957471
Title: A Phase Ia/Ib, Open-Label, First-in-human, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of BC3195 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of BC3195 Monotherapy in Patients With Advanced Solid Tumors
Acronym: BC3195
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocity Biopharmaceutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC3195-101
Record Dates: First submitted 2023-07-13; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BC3195 treatment group. (Experimental): BC3195 via intravenous(IV).
  Interventions: Drug: Drug: BC3195 for Injection

INTERVENTIONS:
Drug: Drug: BC3195 for Injection — BC3195 via intravenous(IV).

SUMMARY:
This is a phase I study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Preliminary Efficacy of BC3195 in Patients with Locally Advanced or Metastatic Solid Tumors.

DETAILED DESCRIPTION:
This is a phase I study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Preliminary Efficacy of BC3195 in Patients with Locally Advanced or Metastatic Solid Tumors.

The patients in whom standard treatment has failed (either due to disease progression or intolerance), who meet the criteria will receive BC3195 via intravenous (IV) in 21-day treatment cycles.

A Safety Monitoring Committee (SMC) will be established to decide the dose levels to be administered and dose regimen during dose escalation based on a thorough review of all the safety, PK (if applicable), and other relevant data from the previous dose cohort, and to determine the MTD and the putative RP2D for dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participate in the study and should provide a written informed consent.
2. Male or female patients ≥ 18 years of age.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Subjects with locally advanced or metastatic solid tumors failed to prior SOCs and no appropriate SOC to treat the current disease per investigator's judgement.
5. Life expectancy ≥ 3 months.
6. Subjects with adequate organ function.
7. Men or women of childbearing potential (which refer to men or women who have not been surgically sterilized and pre-menopausal women) must use a highly effective method of contraception during the study and continue to take contraception measures for 6 months after the last dose of the study drug.

Exclusion Criteria:

1. Pregnant or lactating women.
2. Prior systemic anticancer treatment within 5 half-lives or 4 weeks before the first dose (whichever is shorter).
3. Active viral infection requiring systemic therapy during the screening period.
4. Hypertension that cannot be well-controlled with medical treatment.
5. Cardiovascular disease of clinical significance.
6. Subjects with any active infection that requires anti-infective therapy judged by the investigators.
7. Subjects are not suitable for participating the study judged by the investigators.
8. Subjects with poor compliance, who are unwilling to or unable to follow study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) . | Dose limiting toxicities (DLT) will be assessed At the end of Cycle 1 (each cycle is 21 days).

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China